CLINICAL TRIAL: NCT01213264
Title: Observational Project on the Current Neuromuscular Monitoring Practice (Including Extubation Practice) Via TOF-ratio (Train-of-four) Measurements in Different Types of Surgery After Administration of Neuromuscular Blocking Agents With or Without Reversal (Protocol No. P06556)
Brief Title: Observational Study to Evaluate the Current Neuromuscular Monitoring Practice Used After Different Types of Surgery, for Which Neuromuscular Blocking Agents Were Used, With or Without Blocking Reversal (P06556)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P06556
Record Dates: First submitted 2010-09-09; First posted 2010-10-01 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Neuromuscular Monitoring After Administration of Neuromuscular Blocking Agents in Different Types of Surgery
Keywords: neuromuscular blockade, NMBA, sugammadex, Bridion, TOF,
MeSH Terms: conditions — Tetralogy of Fallot | interventions — Sugammadex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Spontaneous NMB reversal: Participants whose reversal from NMB is spontaneous (no reversal agent used)
  Interventions: Other: No neuromuscular blockade (NMB)-reversal agent used
- NMB reversal with sugammadex: Participants who are administered sugammadex for NMB reversal in accordance with routine anesthesiology practice, and labeling guidelines
  Interventions: Drug: Sugammadex
- NMB reversal with other agents: Participants who are administered any other agent (other than sugammadex) for NMB reversal in accordance with routine anesthesiology practice, and labeling guidelines
  Interventions: Drug: Other NMB-Reversal Agents Used in Routine Anesthesiology Practice

INTERVENTIONS:
Other: No neuromuscular blockade (NMB)-reversal agent used — Participants whose reversal from NMB is spontaneous (no reversal agent used)
  Groups: Spontaneous NMB reversal
Drug: Sugammadex — Participants receive NMB-reversal agents at the discretion of the treating physician per label according to local guidelines, in accordance with routine anesthesiology practice.
  As this is a prospective observational study designed to collect data as part of routine clinical practice, the protocol does not assign which reversal agents, if any, are to be used. This intervention is associated with a cohort that is intended to include participants who receive the NMB-reversal agent sugammadex, administered according to the local clinical practice and drug product labeling.
  Other Names: Bridion; SCH 900616
  Groups: NMB reversal with sugammadex
Drug: Other NMB-Reversal Agents Used in Routine Anesthesiology Practice — Participants receive NMB-reversal agents at the discretion of the treating physician per label according to local guidelines, in accordance with routine anesthesiology practice.
  As this is a prospective observational study designed to collect data as part of routine clinical practice, the protocol does not assign which reversal agents, if any, are to be used. This intervention is associated with a cohort that is intended to include participants who receive any NMB-reversal agent other than sugammadex, and represents multiple drugs whose use and administration may vary according to local clinical practice, product availability and product labeling.
  Groups: NMB reversal with other agents

SUMMARY:
The intent of this observational study is to collect prospective data regarding neuromuscular monitoring practices and extubation standards (Train-Of-Four [TOF] value) during surgery, in countries of Central and Eastern Europe, Middle East and Africa (CEE/EEMEA countries). Secondarily the study will observe, for which surgical procedures neuromuscular blocking agents (NMBAs), and reversal agents to such, are used. This study is a non-interventional clinical trial, and administration of NMBAs, and respective reversal agents, (as well as all drugs used during anesthesia) will be done in accordance with routine anesthesiology practice, and labeling guidelines. Neuromuscular transmission will be monitored according to routine anesthesiology practice by means of acceleromyography. The assignment of the participant to a particular therapeutic strategy is not decided in advance by a trial protocol, but falls within current practice and the prescription of the medicine is clearly separated from the decision to include the patient in the study.

ELIGIBILITY:
Inclusion Criteria

All of the criteria below must be met for a participant to be eligible for study participation.

The prospective participant:

* Is an adult, 18 to 65 years-of-age;
* Is to undergo surgery requiring general anesthesia with non-depolarizing NMBA administration, with or without NMB reversal;
* Meets the inclusion criteria listed on the NMBA label in each country;
* Is willing to participate and sign an informed consent form (ICF).

Exclusion Criteria

Exclusion from the study will be determined by the treating physician. In addition the criteria below should be considered in determining those participants who should be excluded from the study.

The prospective participant:

* Is pregnant or breast feeding;
* Has a neuromuscular disorder;
* Has severe hepatic impairment;
* Has severe renal impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-65 years old) who are undergoing different types of surgical procedures (short, intermediate, or long in duration), requiring general anesthesia with a non-depolarizing NMBA, with or without NMB reversal.
Sampling Method: Non-Probability Sample
Enrollment: 659 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Spontaneous Reversal: Participants whose reversal from neuromuscular blockade (NMB) was spontaneous (no reversal agent used)
- Sugammadex: Participants administered sugammadex for NMB reversal
- Other Reversal Agents: Participants administered any other agent (other than sugammadex) for NMB reversal
Period: Overall Study
Arm/Group | Spontaneous Reversal | Sugammadex | Other Reversal Agents
Started | 155 | 177 | 327
Completed | 153 | 175 | 321
Not Completed | 2 | 2 | 6
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Spontaneous Reversal: Participants whose reversal from NMB was spontaneous (no reversal agent used)
- Total: Total of all reporting groups
Arm/Group | Spontaneous Reversal | Sugammadex | Other Reversal Agents | Total
Number analyzed (Participants) | 155 | 177 | 327 | 659
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (13.7) | 45.3 (13.6) | 42.7 (12.7) | 43.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 106 | 210 | 425
  Male | 46 | 71 | 117 | 234

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Train-Of-Four (TOF)-Ratio <0.9 at Extubation
Description: Neuromuscular function assessment was performed according to routine anesthesiology practice. This typically involves application of repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve and assessment of twitch response at the adductor pollicis muscle. The TOF-ratio, expressed as a decimal from 0.0 up to 1.0, is the ratio of the magnitude of the fourth twitch (T4) to that of the first twitch (T1). The greater the T4/T1 ratio the greater the recovery from neuromuscular blockade. The TOF-ratio was measured at the time of post-surgical extubation. TOF-ratio at time of extubation was to be recorded for each participant, if available, irrespective of the criteria used to make the decision to extubate the participant. TOF-ratio <0.9 at extubation is considered to indicate a high risk for development of postoperative residual curarization (i.e, residual neuromuscular blockade), which can result in respiratory complications.
Time Frame: At extubation (approximately <1 to 125 minutes after end of surgery)
Population: Evaluable participants with TOF-ratio measurement at time of extubation
Measure: Number; unit: participants
Arm/Group | Spontaneous Reversal | Sugammadex | Other Reversal Agents
Number analyzed (Participants) | 137 | 175 | 318
participants | 55 | 17 | 95

2. Primary Outcome: Time From End of Surgery (End of Last Stitch) to Extubation
Description: This measure is the duration from the last surgical wound stitch to the post-surgical extubation of the participant. The time of extubation was to be recorded for each participant, irrespective of the criteria used to make the decision to extubate the participant. Data are presented by TOF-ratio <0.9 and ≥0.9 at extubation. The TOF-ratio is a measure of neuromuscular function ranging from 0.0 to 1.0. The greater the T4/T1 ratio the greater
  the recovery from neuromuscular blockade. TOF-ratio <0.9 at extubation is considered to indicate a high risk for development of postoperative residual curarization (i.e, residual neuromuscular blockade), which can result in respiratory complications.
Time Frame: From end of surgery (end of last stitch) to extubation (duration of approximately <1 to 62 minutes)
Population: Evaluable participants with TOF-ratio measurement at time of extubation and available procedure duration data. Three sugammadex participants with duration from end of surgery to extubation >1 hour were excluded from analysis; delay of extubation was considered due to factors unrelated to administration of sugammadex.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Spontaneous Reversal | Sugammadex | Other Reversal Agents
Number analyzed (Participants) | 137 | 172 | 318
minutes
  TOF-ratio <0.9 at extubation (N=55, 17, 95) | 12.80 (11.54) | 8.82 (5.16) | 11.76 (7.14)
  TOF-ratio ≥0.9 at extubation (N=82, 155, 223) | 9.73 (7.96) | 10.01 (7.28) | 12.20 (6.97)

3. Primary Outcome: Type of Surgical Procedure Performed in Study Participants
Description: The type of surgical procedure performed in each study participant was recorded.
Time Frame: Day of surgery (Day 1)
Population: All study participants who received a neuromuscular blocking agent (NMBA) or NMB-reversal agent
Measure: Number; unit: participants
Groups:
- Total Study Population: Total population of study participants who received an NMBA or NMB-reversal agent
Arm/Group | Total Study Population
Number analyzed (Participants) | 659
participants
  cholecystectomy | 129
  nasal septal operation | 47
  thyroidectomy | 36
  intervertebral disc operation | 34
  hysterectomy | 28
  other surgical procedure | 385

4. Secondary Outcome: Time From NMB-reversal Agent Administration to Operating Room Dismissal
Description: This measure is the duration from NMB-reversal agent administration to dismissal of the participant from the Operating Room. The time of dismissal from the Operating Room was to be recorded for each participant, irrespective of the criteria used to make the decision to dismiss the participant.
Time Frame: Post-surgical period (up to approximately 24 hours post-surgery)
Population: Evaluable participants who received an NMB-reversal agent and had available procedure duration data. Participants in the Spontaneous Reversal group did not receive any NMB-reversal agents and therefore were not included in this analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Other Reversal Agents
Number analyzed (Participants) | 124 | 194
minutes | 15.90 (14.96) | 40.46 (109.9)

5. Secondary Outcome: Time From NMB-reversal Agent Administration to Recovery Room Dismissal
Description: This measure is the duration from NMB-reversal agent administration to dismissal of the participant from the Recovery Room. The time of dismissal from the Recovery Room was to be recorded for each participant, irrespective of the criteria used to make the decision to dismiss the participant.
Time Frame: Post-surgical and recovery period (up to approximately 170 hours post-surgery)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Other Reversal Agents
Number analyzed (Participants) | 130 | 199
minutes | 630.5 (1070) | 619.2 (1348)

6. Primary Outcome: Type of NMB-reversal Agent Administered to Study Participants
Description: For all participants who received an NMB-reversal agent, the specific agent administered was recorded.
Time Frame: At administration of NMB-reversal agent (up to approximately 395 minutes after start of surgery)
Population: All study participants who received an NMBA or NMB-reversal agent
Measure: Number; unit: participants
Arm/Group | Total Study Population
Number analyzed (Participants) | 659
participants
  neostigmine | 327
  sugammadex | 177
  NMB-reversal agent not administered | 155

ADVERSE EVENTS:
Arm/Group | Spontaneous Reversal | Sugammadex | Other Reversal Agents
Serious Adverse Events (participants affected / at risk) | 2/155 | 3/177 | 2/327
Other Adverse Events (participants affected / at risk) | 21/155 | 23/177 | 40/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spontaneous Reversal (N=155) | Sugammadex (N=177) | Other Reversal Agents (N=327)
bradyarrythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Type I hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
airway peak pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
shock haemorrhagic (Vascular disorders) | 2 (3) | 0 (0) | 0 (0)
venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spontaneous Reversal (N=155) | Sugammadex (N=177) | Other Reversal Agents (N=327)
nausea (Gastrointestinal disorders) | 4 (5) | 10 (10) | 10 (10)
procedural pain (Injury, poisoning and procedural complications) | 15 (15) | 14 (14) | 14 (14)
hypotension (Vascular disorders) | 3 (4) | 1 (1) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from Investigator's site will initially only be published/presented with results from the other sites, unless permission is obtained to publish separate results. Investigator will not publish interim results. Sponsor must be able to review all proposed study results communications 45 days prior to submission for publication/presentation. If parties disagree concerning appropriateness of proposed content, Investigator will meet with Sponsor's representatives to discuss/resolve any issues.